CLINICAL TRIAL: NCT06749054
Title: A Phase 2, Open-label, Single-Arm Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Antiviral Activity of Long-Acting Lenacapavir in Combination With an Optimized Background Regimen in Treatment-experienced Adolescents and Children With HIV-1
Brief Title: Evaluation of Long-Acting Lenacapavir for the Treatment of HIV-1 in Treatment-experienced Adolescents and Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-200-6712
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LEN (Experimental): Participants will receive oral LEN 600 mg on Days 1 and 2. Participants will also receive 2 doses of LEN 927 mg as subcutaneous (SC) injection on Day 1 and Week 26 along with their OBR per clinical practice.
  At the Week 52, participants will be given the option to receive SC LEN every 6 months while continuing their OBR for at least another 2 SC LEN doses in the extension phase.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Optimized Background Regimen (OBR)

INTERVENTIONS:
Drug: Oral Lenacapavir — Tablets administered without regard to food
  Other Names: GS-6207; Sunlenca®
Drug: Subcutaneous Lenacapavir — Administered via subcutaneous injections
  Other Names: GS-6207; Sunlenca®
Drug: Optimized Background Regimen (OBR) — Optimized background regimen as prescribed by the Investigator

SUMMARY:
The goal of this clinical study is to learn more about the study drug, lenacapavir (LEN). The study will assess the safety, tolerability, and efficacy of long-acting LEN when combined with other medicines in adolescents and children living with HIV-1 who weigh at least 35 kg and have been treated before for HIV-1. The study will also see how easy it is for participants to take LEN as injection or an oral pill.

The primary objectives are to evaluate the pharmacokinetics and safety of LEN in combination with optimized background regimen (OBR) in TE pediatric participants with HIV-1.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight at screening ≥ 35 kg.
* On a stable failing antiretroviral (ARV) regimen for > 8 weeks before screening and willing to continue the regimen until Day 1.
* Plasma HIV-1 RNA ≥ 400 copies/mL on at least 2 consecutive occasions spanning at least 6 months, including at screening.
* Have previously changed their ARV regimen due to treatment failure.
* ARV treatment options limited due to resistance, tolerability, contraindications, safety, drug access.
* Able and willing to commit to taking LEN in combination with their OBR.
* The following laboratory parameters at screening:

  1. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m^2 using Bedside Schwartz Formula.
  2. Absolute neutrophil count > 0.50 GI/L (> 500 cells/mm^3).
  3. Hemoglobin ≥ 85 g/L (> 8.5 g/dL).
  4. Platelets ≥ 50 GI/L (≥ 50,000/mm^3).
  5. Hepatic transaminases (aspartate aminotransferase and alanine aminotransferase) ≤ 5 × upper limit of normal.
  6. Total bilirubin ≤ 23 μmol/L (≤ 1.5 mg/dL) and direct bilirubin ≤ 7 μmol/L (≤ 0.4 mg/dL).

Key Exclusion Criteria:

* Life expectancy ≤ 1 year.
* An opportunistic illness requiring treatment within the 30 days prior to screening.
* Evidence of active pulmonary or extra-pulmonary tuberculosis within 3 months prior to screening.
* Hepatitis C virus (HCV) antibody positive with detectable HCV RNA at screening.
* Hepatitis B virus (HBV) surface antigen (HBsAg) positive or HBV core antibody (antibody against hepatitis B core antigen (anti-HBc)) positive; if individual is HBsAg negative and anti-HBc positive but HBV DNA undetectable, individual may be enrolled.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Ctrough, W26 of Lenacapavir (LEN) | Week 26
  Ctrough, W26 is defined as the plasma concentration at the end of the dosing interval at Week 26.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events (AEs) Through Week 26 | First dose date up to Week 26
Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Through Week 26 | First dose date up to Week 26

SECONDARY OUTCOMES:
PK Parameter: Cmax, D1-W26 of LEN | Day 1 up to Week 26
  Cmax, D1-W26 is defined as the maximum observed concentration of drug from Day 1 to Week 26.
PK Parameter: AUC D1-W26 of LEN | Day 1 up to Week 26
  AUC D1-W26 is defined as the partial area under the concentration versus time curve from Day 1 to Week 26.
Percentage of Participants Experiencing Treatment-Emergent AEs Through Week 52 | First dose date up to Week 52
Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Through Week 52 | First dose date up to Week 52
Percentage of Participants With Plasma HIV-1 RNA < 50 Copies/mL at Week 26 Based on the US Food and Drug Administration (FDA)-Defined Snapshot Algorithm | Week 26
Percentage of Participants with Plasma HIV-1 RNA < 50 Copies/mL at Week 52 Based on the US FDA-Defined Snapshot Algorithm | Week 52
Change From Baseline in Clusters of Differentiation (CD4)+ Cell Counts at Week 26 | Baseline, Week 26
Change From Baseline in CD4+ Cell Counts at Week 52 | Baseline, Week 52
Percent Change From Baseline in CD4+ at Week 26 | Baseline, Week 26
Percent Change From Baseline in CD4+ at Week 52 | Baseline, Week 52
General Acceptability of Oral LEN as Assessed by Percentage of Participants With Acceptability Questionnaire Responses on Day 1 | Day 1
  To assess the acceptability of the study drug, the participants will complete questionnaire including a question on general acceptability of the assigned study drug on an ordinal 5-category scale.
General Acceptability of Oral LEN as Assessed by Percentage of Participants With Acceptability Questionnaire Responses on Day 2 | Day 2
  To assess the acceptability of the study drug, the participants will complete questionnaire including a question on general acceptability of the assigned study drug on an ordinal 5-category scale.
General Palatability of Oral LEN as Assessed by Percentage of Participants With Palatability Questionnaire Responses on Day 1 | Day 1
  To assess the palatability of the study drug, the participants will complete questionnaire including a question on general palatability of the assigned study drug on an ordinal 5-category scale.
General Palatability of Oral LEN as Assessed by Percentage of Participants With Palatability Questionnaire Responses on Day 2 | Day 2
  To assess the palatability of the study drug, the participants will complete questionnaire including a question on general palatability of the assigned study drug on an ordinal 5-category scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- Grady Health System, Ponce De Leon Center, Atlanta, Georgia, United States
- South Africa (8):
  - FAMCRU, Cape Town
  - CRISMO Research Centre, Germiston
  - Wits RHI Shandukani Research Centre CRS, Johannesburg
  - Rahima Moosa Mother and Child Hospital, Johannesburg
  - Clinical Research Institute of South Africa (CRISA), KwaDukuza
  - Durban International Clinical Research Site, Enhancing Care Foundation, KwaZulu - Natal
  - Be Part Research Pty (Ltd), Paarl
  - Perinatal HIV Research Unit (PHRU), Soweto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06749054